CLINICAL TRIAL: NCT00347724
Title: Double-blind, Randomized, Placebo-controlled, Parallel Group Comparison of the Efficacy and Safety of Extended Release Tramadol (Tramadol ER) 300 mg and 200 mg to Placebo in the Treatment of Chronic Low Back Pain
Brief Title: A Study Comparing the Effectiveness and Safety of Extended-release Tramadol Versus Placebo in the Treatment of Chronic Low Back Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bausch Health Americas, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: B00.CT3.014.TRA P03
Record Dates: First submitted 2006-07-02; First posted 2006-07-04 (Estimated); Last update posted 2012-06-21 (Estimated); Status verified 2012-06

CONDITIONS: Chronic Pain
Keywords: chronic low back pain; chronic pain; low back pain; extended-release analgesia; opioid
MeSH Terms: conditions — Chronic Pain; Low Back Pain

INTERVENTIONS:
Drug: Tramadol HCl ER

SUMMARY:
The purpose of this study is to compare the analgesic efficacy of oral, once-daily tramadol ER 300 mg and 200 mg to placebo in patients with moderate to severe chronic low back pain requiring daily analgesic treatment. The study hypothesis is that tramadol ER is effective in the treatment of moderate to severe chronic low back pain.

DETAILED DESCRIPTION:
Immediate release (IR) tramadol has demonstrated efficacy in several pain conditions including: obstetrical, gynecological, orthopedic, abdominal, and oral surgery. The short elimination half-life of IR tramadol necessitates every 4-6 hour dosing in order to maintain optimum levels of analgesia in chronic pain. The study medication in this study is a once-daily, extended release (ER) tramadol formulation. This is a multicenter, double-blind, randomized, placebo-controlled, parallel-group study. At the Screening Visit, patients eligible for study participation by medical history, physical exam and other evaluations will enter a 2-7 day washout period during which time analgesics will not be allowed. At Visit 2, patients with a pain intensity >= 40 mm on a 100 mm visual analog scale (VAS) and who meet all other eligibility criteria will be admitted into a 3-week, open-label, run-in period during which time they will receive tramadol ER 100 mg once daily (QD) for at least 3 days. On Day 4, the dose will be increased to tramadol ER 200 mg QD, based on tolerability. Patients must be maintained on a minimum dose of tramadol 200 mg QD by the beginning of Week-2 (Visit 3); the dose may be increased to tramadol ER 300 mg QD at Visit 3, based on tolerability. Patients must increase their tramadol ER dose to 300 QD by the beginning of Week - 1 (Visit 4); this dose must be maintained for one week. Patients with pain unresponsive to appropriate dose adjustments or with unacceptable side effects will be discontinued from the study and an alternative analgesic therapy will be initiated. Patients receiving tramadol ER 300 mg QD at the end of the run-in period (Visit 5, Week 0) will enter a 12-week, double-blind period during which they will be randomized to receive tramadol ER 300 mg, tramadol ER 200 mg, or placebo QD. No dose adjustments will be permitted during the double-blind period of the study. Patients will return for safety and efficacy evaluations at Weeks 1, 2, 4, 8 and 12 or early termination. Study medication will be discontinued at Week 12 and patients will return after one week for a post-treatment visit (Week 13).

ELIGIBILITY:
Inclusion Criteria:

* Patients with a history of chronic low back pain >= 6 months requiring treatment with NSAIDs, acetaminophen, opioid analgesics, COX-2 selective inhibitors, and/or muscle relaxants for at least 60 of the 90 days preceeding the screening visit; in good health as determined by the investigator on the basis of medical history, physical exam and screening labs; patient's low back pain intensity measures >= 40 mm on a visual analog scale (VAS) at the start of the run-in peroid after the 2-7 day washout; patients who are able to discontinue treatment with NSAIDs, COX-2 selective inhibitors, tramadol, muscle relaxants, opioids, and/or other analgesics during the 2-7 day washout period and all other analgesics throughout the entire study.

Exclusion Criteria:

* Patients with a diagnosis of a complex regional pain syndrome, significant inflammatory pain, or clinically significant active fibromyalgia; patients with a history of lumbar surgery or chemonucleolysis; patients undergoing transcutaneous electrical nerve stimulation (TENS) or spinal manipulation for low back pain; patients with an uncontrolled medical condition or a clinically significant condition that would, in the investigator's opinion, preclude study participation; patients using analgesics or other agents during washout that could confound the analgesic response.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600
Dates: Start 2000-11; Study Completion 2001-11

PRIMARY OUTCOMES:
Patient's pain intensity score since the previous visit,using a visual analog scale(VAS) where 0 mm = no pain and 100 mm = extreme pain.

SECONDARY OUTCOMES:
Patient's current pain intensity VAS score
Patient's global assessment
Roland Disability Index
Patient's sleep assessment